CLINICAL TRIAL: NCT02119312
Title: General Screening for Eligibility to Participate in Treatment, Prevention and Vaccine Trials at the Seattle Malaria Clinical Trials Center
Brief Title: Malaria Clinical Trials Center General Screening
Acronym: GS
Status: Completed | Type: Observational
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: MC-002
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Malaria
Keywords: Malaria; Plasmodium; Plasmodium falciparum; Clinical Trials; Vaccine Study; Drug Study; Malaria Clinical Trials Center; Seattle BioMed; Center for Infectious Disease Research
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to identify and screen potential subjects for preliminary eligibility to participate in a malaria related clinical trial conducted at the Seattle Malaria Clinical Trials Center (Seattle MCTC) or one of our partnering sites.

DETAILED DESCRIPTION:
This is a continuous study enrolling approximately 350 participants per year to establish preliminary eligibility for participation in ongoing or future Seattle Malaria Clinical Trials Center (Seattle MCTC) clinical research studies. Data collected may be used to support preliminary eligibility for a current or future Seattle MCTC clinical research study.

In order to maximize efficiency of the screening process potential participants who contact the site will be pre-screened using an IRB-approved screening form.

Potential participants who contact the site may be asked to come in for an in-person screening visit. They will be given a consent form to read and sign if they should choose to participate in the screening process. If they have any questions during this process research staff will be available. This visit includes an in-depth medical history review, travel history, physical exam, blood draw, electrocardiogram test (ECG), and a urine test.

The Seattle Malaria Clinical Trials Center (Seattle MCTC) is conducting research to combat malaria. Malaria is a disease that is transmitted to humans by the bite of an infected mosquito and affects millions of people worldwide. Malaria can cause a wide range of medical problems, and may even result in death if the infection is not treated. Currently there are many medications, preventative measures and malaria vaccines being developed to fight malaria that will need to be tested before they can be made available to the general public. The Seattle MCTC is conducting clinical research studies for this purpose and is in need of healthy adult volunteers to take part in upcoming studies.

ELIGIBILITY:
Inclusion Criteria:

* Good general health status as demonstrated by medical history, physical exam, and screening laboratory tests;
* No history of certain chronic medical illnesses (e.g. diabetes, epilepsy, autoimmune disease, hepatitis, heart disease);
* HIV, Hepatitis B and C negative;
* Low risk for coronary heart disease;
* Ability and willingness to provide informed consent;
* Reliable access to the MCTC and associated sites; and
* If participant is biologically female she must not be pregnant and must agree to consistently use an effective form of birth control 21 days prior to enrollment in an active clinical study and for the duration of that study.

Exclusion Criteria:

* Prior receipt of an investigational malaria vaccine;
* Chronic use of systemic antibiotics or immunosuppressive medications with anti-malarial effects;
* Chronic medical condition, physical examination findings, other clinically significant abnormal laboratory results, or past medical history that may have clinically significant implications for current health status;
* History of systemic anaphylaxis;
* History of, or known active cardiac disease;
* Elevated (moderate of high) risk of coronary heart disease;
* Clinically significant ECG findings;
* Chronic or active neurological disease;
* History of splenectomy or functional asplenia;
* History of psoriasis or porphyria;
* History of diagnosed ocular disease;
* Positive history of HIV, Hepatitis B and/or C;
* Pregnant or lactating females or females who intend to become pregnant during study period;
* Certain psychiatric conditions that could affect study compliance; and
* Suspected or known current alcohol and/or drug abuse.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Men and non-pregnant women who are in general good health.
Sampling Method: Probability Sample
Enrollment: 2101 (Actual)
Dates: Start 2010-06; Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Participant Enrollment | Once upon enrollment
  See inclusion/exclusion criteria.

CONTACTS AND LOCATIONS:
Overall Officials: James G Kublin, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- See also: Seattle Malaria Clinical Trials Center — http://www.seattlemalaria.org